CLINICAL TRIAL: NCT02567760
Title: Development and Evaluation of a Cognitive Enhancement Product Made From Selected Thai Herbs for Menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jintanaporn Wattanathorn, Associated Professor Doctor, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HE 571329
Record Dates: First submitted 2015-09-18; First posted 2015-10-05 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: MP1; cognitive enhancing effect; menopausal women

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MP1 group (Active Comparator): Subjects receive the MP1 product at the dose of 400 mg/day for 8 weeks.
  Interventions: Dietary Supplement: MP1
- Placebo group (Placebo Comparator): Subject receive the Placebo product for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MP1 — Subjects receive MP1 drink at the dose of 400 mg/day after meal for 8 weeks.
  Arms: MP1 group
Other: Placebo — Subjects receive Placebo drink after meal for 8 weeks.
  Arms: Placebo group

SUMMARY:
This study is set up to determine the cognitive enhancing effect and consumption safety of the novel cognitive enhancement product made from the combined extract of Z. mays (purple color) and P. amaryllifolius based-drink (MP1) in menopausal volunteer.

DETAILED DESCRIPTION:
Memory impairment is one of the common health problems in menopausal women. Due to the therapeutic efficiency limitation, the searching for the protective intervention for this condition is required. Based on the previous findings that the combined extract of Z. mays (purple color) and P. amaryllifolius based-drink (MP1) could attenuate memory impairment in animal model of menopause, the investigators aimed to investigate the effect of MP1 functional drink on working memory, psychological fitness, possible underlying mechanism and the consumption safety in menopausal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy perimenopausal and postmenopausal women (<5 years menstruation cessation) who live in Northeastern of Thailand.

Exclusion Criteria:

* Subject who is diagnosed with one of the following: cardiovascular diseases, respiratory diseases,neuropsychological diseases, head injury, diabetes mellitus, liver disease, cancer, autoimmune disease and hematological disorder are excluded.
* Hysterectomy and/or Oophorectomy
* Subject who use hormone or any drug exerts the influence on Hypothalamic Pituitary Gonadal axis and nervous system.
* Body mass index >27
* Athlete or subject who has a regular exercise.
* Smoker or heavy drinker

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cognitive processing (P300) and attention (N100) using Event Related Potential | 7 months

SECONDARY OUTCOMES:
Accuracy and speed of working memory using computerized battery test | 7 months
Psychological fitness using Bond-Ladder test and Symptom Check List-90 test (SCL-90) | 7 months
Malondialdehyde level in serum | 7 month
The activity of Superoxide dismutase enzyme in serum | 7 month
  The activity of Superoxide dismutase (SOD) enzyme in serum is measured by using the biochemical assay method and the activity of SOD is expressed as units/mg protein. The higher activity of SOD enzyme is the better antioxidant effect of the intervention.
The activity of Glutathione Peroxidase enzyme in serum | 7 month
  The activity of Glutathione Peroxidase (GSH-Px) enzyme in serum is measured by using the biochemical assay method and the activity of GSH-Px is expressed as units/mg protein. The higher activity of GSH-Px enzyme is the better antioxidant effect of the intervention.
The activity of Catalase enzyme in serum | 7 month
  The activity of Catalase enzyme in serum is measured by using the biochemical assay method and the activity of CAT is expressed as units/mg protein. The higher activity of CAT enzyme is the better antioxidant effect of the intervention.
The activity of Acetylcholinesterase enzyme in serum | 7 month
  Acetylcholinesterase (AChE) is an enzyme that catalyzes the breakdown of Acetylcholine, a neurotransmitter for learning and memory.The activity of AChE enzyme in serum is measured by using the biochemical assay method and the result is express as mmol/min.g protein. The lower activity of AChE is the better cognitive enhancing effect of the intervention.
The activity of Monoamine oxidase enzyme in serum | 7 month
  Monoamine oxidase (MAO) is an enzyme that catalyzes the breakdown of Monoamine neurotransmitter , a neurotransmitter for learning and memory.The activity of MAO enzyme in serum is measured by using the biochemical assay method and the result is express as nmol/h/mg protein. The lower activity of MAO is the better cognitive enhancing effect of the intervention.
Consumption safety of MP1 by using the electrocardiogram (ECG), Blood chemistry, hematology, blood pressure measurement | 7 months
Adverse events by using adverse event record form | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Jintanaporn Wattanathorn, PhD, Principal Investigator — Khon Kaen University